CLINICAL TRIAL: NCT02672644
Title: A Single-Center, Non-Comparative Study to Evaluate Subject Recovery Following Correction of Bilateral Nasolabial Folds Using Emervel® Classic Lidocaine and Emervel® Deep Lidocaine
Brief Title: Non-comparative Evaluation of Facial Expressions Following Lower Face Correction Using Emervel Classic and Emervel Deep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10346
Record Dates: First submitted 2016-01-26; First posted 2016-02-03 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2016-07

CONDITIONS: Nasolabial Folds; Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Emervel Classic (Experimental): Subjects treated with Emervel Classic (moderate NLFs; WSRS = 3/3). Subjects receiving bilateral treatment of NLFs following approved product labeling.
  Interventions: Device: Emervel Classic
- Emervel Deep (Experimental): Subjects treated with Emervel Deep (severe NLFs; WSRS = 4/4). Subjects receiving bilateral treatment of NLFs following approved product labeling.
  Interventions: Device: Emervel Deep

INTERVENTIONS:
Device: Emervel Classic — Subjects requiring bilateral correction of NLFs and meeting eligibility criteria will be enrolled and treated with Emervel Classic (moderate NLFs; WSRS = 3/3)
  Arms: Emervel Classic
Device: Emervel Deep — Subjects requiring bilateral correction of NLFs and meeting eligibility criteria will be enrolled and treated with Emervel Deep (severe NLFs; WSRS = 4/4).
  Arms: Emervel Deep

SUMMARY:
Study is designed to characterize subject and treating investigator reported outcomes in the early post-treatment period, following bilateral correction of nasolabial folds using Emervel Classic and Emervel Deep.

1. to evaluate subject-reported return to social engagement, after the initial treatment (Baseline/Day 1 visit).
2. to evaluate change in Global Aesthetic Improvement Scale (GAIS) at day 30- subject/investigator reported
3. to evaluate subject satisfaction with treatment outcome at baseline, day 14 and day 30.
4. to evaluate change in Wrinkle Severity Rating Scale (WSRS) from baseline to post-treatment follow-up time points at day 14 and Day 30 - investigator reported
5. to evaluate all adverse events during the course of the study

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subjects, 35 to 60 years of age
2. Bilateral NLFs: severe (WSRS = 4/4) or moderate (WSRS = 3/3), as assessed by the treating investigator
3. Subjects of childbearing potential who agree to use medically accepted methods of contraception during the study and for 30 days following study completion.

Childbearing potential is defined as not being surgically sterile (e.g., hysterectomy, bilateral salpingo-oophorectomy, or tubal ligation) or those who are not post-menopausal (absence of menstruation for at least 1 year prior to Day 1).

- If not surgically sterile or post-menopausal, the subject agrees to use acceptable forms of contraception. Acceptable methods of contraception are defined as follows:

1. use of oral/systemic contraceptives for at least 3 months prior to the start of the study; or
2. use of an intrauterine device; or
3. use of double barrier (e.g., condom or diaphragm and spermicidal foam/gel, condom and diaphragm); or
4. use of contraceptive implants or injectables for at least 28 days prior to the start of the study; or
5. partner with vasectomy at least 3 months prior to study start; or
6. strict abstinence.

Females of child bearing potential must have negative urine pregnancy test (UPT) at Day 1 and Day 14 if touch-up is to be performed.

Key Exclusion Criteria:

1. Subject who presents with a severity of wrinkles or folds that require other treatments, e.g. laser treatment, chemical peeling, to achieve optimal correction
2. Previous facial surgery, including aesthetic facial surgical therapy, liposuction or tattoo, in the treatment area
3. Previous tissue augmenting therapy or contouring with permanent filler-type injectable product
4. Previous tissue augmenting therapy with non-permanent filler or fat-injection in the facial area to be treated, within twelve (12) months before treatment
5. Previous tissue revitalisation treatment with neurotoxin below the zygomatic arch, within six (6) months before treatment
6. Previous tissue revitalisation treatment with laser or light, mesotherapy, chemical peeling or dermabrasion below the zygomatic arch within six (6) months before treatment
7. Subject who presents with severe midface volume loss
8. Subject has a beard or facial hair that, in the investigator's opinion, would interfere with the study injections and/or study assessments
9. Woman who plans to become pregnant during the study
10. Woman who is pregnant or breast feeding
11. Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel
12. Known/previous allergy or hypersensitivity to local anaesthetics, e.g. lidocaine or other amide-type anaesthetics
13. Known/previous allergy or hypersensitivity to gram-positive bacterial proteins
14. History of severe or multiple allergies manifested by anaphylaxis
15. History of bleeding disorders or treatment with anticoagulants or inhibitors of platelet aggregation within two (2) weeks before treatment
16. Treatment with chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic or topical (facial) corticosteroids (inhaled corticoids are allowed) within three (3) months before study treatment
17. Any medical condition or treatment that, in the opinion of the treating investigator, would make the subject unsuitable for inclusion
18. Study site personnel, close relatives of the study site personnel (e.g. parents, children, siblings, or spouse), employees, or close relatives of employees at the Sponsor company
19. Participation in any clinical study within thirty (30) days before treatment

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Subject-reported time of return to social engagement after initial treatment | 30 days
  Time of return to social engagement (in hours)

SECONDARY OUTCOMES:
Change from baseline to post-treatment follow-up time points in subject reported GAIS | up to 30 days
  Change from baseline to post-treatment follow-up time points in the subject reported GAIS (photographs) at day 30
Subject satisfaction with treatment outcome of the nasolabial folds | 30 days
  Subject satisfaction with treatment assessments at baseline, day 14, and day 30
Change from baseline to post-treatment follow-up time points in treating investigator reported WSRS | 30 days
  Change from baseline to post-treatment follow-up time points in the treating investigator reported WSRS at day 14 and day 30
Change from baseline to post-treatment follow-up time points in treating investigator reported GAIS | 30 days
  Change from baseline to post-treatment follow-up time points in the treating investigator reported GAIS (photographs) at day 30
Incidence rate of subjects with adverse events (AEs) | 30 days
Incidence rate of subjects with injection-related adverse events | 30 days
  Injection-related adverse events recorded by the subject in study diary

CONTACTS AND LOCATIONS:
Overall Officials: Author Swift, MD, Principal Investigator — Arthur Swift Research Inc
Locations (1):
- Arthur Swift Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No